CLINICAL TRIAL: NCT06915571
Title: Assessment of Ankle Mobility, Flexibility, and Y-Balance Test Before and After Plantar Fascia Stretching and Plantar Fascia Stretching Combined With Graston Technique in Recreationally Active Young Adults: A Randomized Controlled Study
Brief Title: The Effect of Graston Technique on Ankle Mobility, Sit-Reach Test and Y-Balance Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, Assistant Professor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-576; Academician (Other: University of Health Sciences Türkiye)
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Plantar Fascia; Flexibility; Y-balance Performance; Recreational Activities; Exercise
Keywords: plantar fascia; flexibility; y-balance performance; recreactional activities; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: One group will undergo plantar fascia stretching. In the other group, graston technique will be applied in addition to plantar fascia stretching. Participants in the study will be between the ages of 18-35.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plantar Fascia Stretching. (Experimental): In the sitting and cross-legged position, the patient will be taught self-plantar fascia stretching. It will be done with 10 repetitions for each 2 extremities.
  Interventions: Other: Plantar Fascia Stretching.
- Plantar Fascia Stretching and Graston Technique Application (Experimental): The patient will be taught self-plantar fascia stretching in sitting and cross-legged position. It will be done with 10 repetitions for each 2 extremities. Then, in prone position, 5 minutes of Graston application will be performed on both plantar fascia.
  Interventions: Other: Plantar Fascia Stretching.; Other: Graston Technique

INTERVENTIONS:
Other: Plantar Fascia Stretching. — It consists of participants who will undergo plantar fascia stretching.
Other: Graston Technique — It consists of participants who will underwent graston technique application.
  Arms: Plantar Fascia Stretching and Graston Technique Application

SUMMARY:
This study investigates the effects of plantar fascia stretching and plantar fascia stretching with graston application on ankle mobility, flexibility and Y-Balance test results in recreationally active young adults. By comparing the effects of the two treatment methods on ankle function, it aims to demonstrate the potential benefits of both treatments.

It was intended to involve 60 participants, or 95% of the interval 0.80's study power.

DETAILED DESCRIPTION:
The plantar fascia, also known as the plantar aponeurosis, is a thick, fibrous band of connective tissue that extends from the medial tubercle of the calcaneus to the proximal phalanges of the toes. It consists of three different segments: medial, central and lateral bands.

The Graston technique (GT) is an instrument-assisted soft tissue mobilization technique that reduces pain, improves overall function and increases range of motion. GT reduces the overall rehabilitation time, uses less pressure and energy, and increases the depth of tissue that can be treated. Furthermore, GT does not compress tissues; the superficial fascia layer is easily mobilized, allowing access to deeper restrictions.

The Y-Balance Test (YBT) is a clinical measurement tool used to assess dynamic balance. Asymmetries between extremities in the anterior direction have been associated with a 2-fold increased risk of lower extremity injury. This study examines how ankle mobility, flexibility, and Y-Balance examination results are affected in young adults who engage in recreational activities by plantar fascia stretching and plantar fascia stretching with graston application. It seeks to illustrate the possible advantages of both therapies by contrasting how the two approaches affect ankle function. People between the ages of 18 and 35 who regularly exercise for leisure at least two to three times a week and who have signed a voluntary permission form committing to actively participate in all study phases will be included. If a participant has a history of lower limb, plantar fascia, or ankle injuries, has had a major injury, surgery, or trauma to the lower extremities in the previous six months, plays professional sports, or declines to participate or withdraws during the evaluations, they will be disqualified. The control group will receive plantar fascia stretching. In addition to stretching the plantar fascia, the experimental group will also receive graston method treatment. A goniometer will be used to objectively measure ankle mobility both before and after the treatment. The Sit and Reach Box (Lafayette Instrument Sit and Reach Box, Flexibility Tester) at the faculty will be used to measure the applicant's flexibility both before and after the application. The participants' balance will be evaluated using the Y Balance TestTM. There shouldn't be any risks or difficulties prior to, during, or following the tests and procedures. It was intended to involve 60 participants, or 95% of the interval 0.80's study power.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-35
* Doing regular physical activity at least 2-3 times a week (Individuals who do sports recreationally)
* Individuals who signed the voluntary consent form before participating in the study and agreed to participate in all stages consciously

Exclusion Criteria:

* Having an ankle injury, plantar fascia or lower limb condition
* Serious injury, surgery or trauma to the lower extremity within the last 6 months
* Individuals practicing sports at a professional level
* Not volunteering to participate in the study or wanting to leave the study during the assessments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Ankle Mobility | before and after the intervention, within 1 hour
  Ankle mobility; dorsiflexion, plantar flexion, inversion and eversion movements will be evaluated with a goniometer before and after the intervention.
Flexibility Assessment | before and after the intervention, within 1 hour.
  Flexibility Assessment, Sit and Reach Test will be measured before and after the intervention using the Flexibility Measurement Stand
Balance | before and after the intervention, within 1 hour.
  Balance assessment will be measured before and after the intervention with the Y-Balance test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Venosa M, Romanini E, Vitale L, Logroscino G. Spontaneous rupture of the plantar fascia: a case report. Front Rehabil Sci. 2024 Aug 27;5:1470002. doi: 10.3389/fresc.2024.1470002. eCollection 2024. PMID 39257473
- [Background] DiGiovanni BF, Nawoczenski DA, Lintal ME, Moore EA, Murray JC, Wilding GE, Baumhauer JF. Tissue-specific plantar fascia-stretching exercise enhances outcomes in patients with chronic heel pain. A prospective, randomized study. J Bone Joint Surg Am. 2003 Jul;85(7):1270-7. doi: 10.2106/00004623-200307000-00013. PMID 12851352
- [Background] Hartley EM, Hoch MC, Boling MC. Y-balance test performance and BMI are associated with ankle sprain injury in collegiate male athletes. J Sci Med Sport. 2018 Jul;21(7):676-680. doi: 10.1016/j.jsams.2017.10.014. Epub 2017 Nov 6. PMID 29102301
- [Background] Bergevin MA, Daugherty CC, Bove KE, McAdams AJ. The internal carotid artery siphon in children and adolescents. Hum Pathol. 1991 Jun;22(6):603-6. doi: 10.1016/0046-8177(91)90239-l. PMID 1864591
- [Background] Abdel-Aal NM, Elsayyad MM, Megahed AA. Short-term effect of adding Graston technique to exercise program in treatment of patients with cervicogenic headache: a single-blinded, randomized controlled trial. Eur J Phys Rehabil Med. 2021 Oct;57(5):758-766. doi: 10.23736/S1973-9087.21.06595-3. Epub 2021 May 5. PMID 33947825